CLINICAL TRIAL: NCT05719363
Title: Portable Oxygen Concentrator in Non-hospitalized Patients With Chronic Heart Failure: A Proof-of-concept Pilot Study
Brief Title: Portable Oxygen Concentrator in Non-hospitalized Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: INO-03
Record Dates: First submitted 2023-01-25; First posted 2023-02-09 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Masking Description: All patients will have the nasal cannula in place during both 6MWTs, but the POC will be activated only during the test conducted with oxygen supplementation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- POC ON (Experimental): 6MWT with Inogen Rove 6 POC turned ON
  Interventions: Device: Inogen Rove 6 Portable Oxygen Concentrator
- POC OFF (Sham Comparator): 6MWT with Inogen Rove 6 POC turned OFF
  Interventions: Device: Inogen Rove 6 Portable Oxygen Concentrator

INTERVENTIONS:
Device: Inogen Rove 6 Portable Oxygen Concentrator — The Inogen Rove 6 POC is designed to provide a flow of high-purity oxygen. Inogen Rove 6 is a highly versatile and robust concentrator which offers patients the option to use up to 6 different flow settings.
  The unit weighs just under 5 pounds. Utilizing an Intelligent delivery technology, the unit can provide patients with required oxygen therapy on a 24/7 basis. The Inogen Rove 6 POC will be used for patients with chronic heart failure as an investigational device. It supplies a high concentration of oxygen and is used with a nasal cannula which channels oxygen from the concentrator to the patient.

SUMMARY:
This is a one-day, proof-of-concept, pilot study of portable oxygen concentrator (POC) administration and Six Minute Walk Test (6MWT) distance in patients with stable chronic heart failure.

DETAILED DESCRIPTION:
This is a one-day, proof-of-concept, pilot study of portable oxygen concentrator (POC) administration and Six Minute Walk Test (6MWT) distance in patients with stable chronic heart failure. A total of 20 patients will be enrolled and undergo two 6MWT on the same day, with Inogen Rove 6 POC turned ON and turned OFF. They will be randomly assigned in a 1:1 ratio to either perform the first 6MWT with Inogen Rove 6 POC turned ON and the second 6MWT with Inogen Rove 6 POC turned OFF, or vice-versa (first and second 6MWT with Inogen Rove 6 POC turned OFF and turned ON, respectively).

Study Description: This is a one-day, proof-of-concept, pilot study of portable oxygen concentrator (POC) administration and Six Minute Walk Test (6MWT) distance in patients with stable chronic heart failure. A total of 20 patients will be enrolled and undergo two 6MWT on the same day, with Inogen Rove 6 POC turned ON and turned OFF. They will be randomly assigned in a 1:1 ratio to either perform the first 6MWT with Inogen Rove 6POC turned ON and the second 6MWT with Inogen Rove 6 POC turned OFF, or vice-versa (first and second 6MWT with Inogen Rove 6 POC turned OFF and turned ON, respectively).

On the day of the only study visit, informed consent will be obtained, inclusion/exclusion criteria will be assessed, and the following information will be obtained: patient demographics, cardiovascular medical history (including heart failure history), NYHA score, heart failure history, respiratory condition history, smoking history, review of current heart failure medications and other cardiovascular concomitant medications.

Eligible patients will be randomly assigned (in a 1:1 ratio) to one of the following 2 sequences:

1. first 6MWT with Inogen Rove 6 POC turned ON followed by a second 6MWT with the Inogen Rove 6 POC turned OFF, or
2. first 6MWT with the Inogen Rove 6 POC turned OFF, followed by a second 6MWT with the Inogen Rove 6 POC turned ON.

There will be a resting period of 60 minutes between the 2 walking tests. POC administration will be started 15 minutes prior to the 6MWT.

The following assessments/procedures will be done:

* 6MWT distance
* Peripheral oxygen saturation on fingertip pulse oximetry before the 6MWT, at 3 minutes (middle of the 6MWT), 6 minutes (end of the 6MWT), and 9 minutes (3 minutes after the end of the 6MWT)
* Heart rate before the 6MWT, at 3 minutes (middle of the 6MWT), at 6 minutes (end of the 6MWT), and at 9 minutes (3 minutes after the end of the 6MWT)
* Modified Borg Scale (5) assessed before the 6MWT, at 3 minutes (middle of the 6MWT), 6 minutes (end of the 6MWT), and 9 minutes (3 minutes after the end of the 6MWT) Safety will be assessed by the monitoring of adverse events (AEs) and serious adverse events (SAEs) related to the use of the POC as well as by evaluating the tolerance to the use of the POC during exercise (ability to complete the 6MWT with the POC).

Objectives:

Main objectives:

To describe the effect of the Inogen Rove 6 POC on:

* 6MWT
* Oxygen saturation level on fingertip pulse oximetry collected before and at 3 minutes (middle of the 6MWT), at 6 minutes (end of the 6MWT), and at 9 minutes (3 minutes after the end of the 6MWT)
* Heart rate before and at 3 minutes (middle of the 6MWT), at 6 minutes (end of the 6MWT), and at 9 minutes (3 minutes after the end of the 6MWT)
* Modified Borg Scale collected before and at 3 minutes (middle of the 6MWT), at 6 minutes (end of the 6MWT), and at 9 minutes (3 minutes after the end of the 6MWT)

Other objectives:

To describe the effect of the Inogen Rove 6 POC on:

* Safety of the Inogen Rove 6 POC in this subject population
* Tolerance to use of the POC during exercise

Endpoints: Main endpoints:

* Walking distance during the 6MWT
* Oxygen saturation on fingertip pulse oximetry at 3 minutes (middle of the 6MWT), at 6 minutes (end of the 6MWT), and at 9 minutes (3 minutes after the end of the 6MWT)
* Heart rate at 3 minutes (middle of the 6MWT), at 6 minutes (end of the 6MWT), and at 9 minutes (3 minutes after the end of the 6MWT)
* Modified Borg Scale at 3 minutes (middle of the 6MWT), at 6 minutes (end of the 6MWT), and at 9 minutes (3 minutes after the end of the 6MWT)

Other endpoints:

* Adverse events (AEs) and serious adverse events (SAEs)
* Ability to complete the 6MWT using the POC

Study Population: Inclusion criteria (all need to be met):

1. Adult male or female
2. Diagnosed with chronic stable heart failure
3. NYHA functional class II to ambulatory class IV
4. Peripheral oxygen saturation on fingertip pulse oximetry (SpO2) ≤96% at rest
5. Willingness and ability to use a POC and with no allergy to cannula material
6. Patient with the capacity to provide informed consent

Exclusion criteria (no exclusion criterion should be met):

1. Contraindication to the use of POC
2. Patient currently hospitalized or requiring hospitalization
3. Current acute decompensated HF requiring augmented therapy with vasodilator agents, and/or inotropic drugs, and/or augmented therapy or i.v. therapy with diuretics
4. History of acute coronary syndrome (unstable angina or myocardial infarction) within 3 months prior to study enrollment
5. Patient unable to walk
6. Patient who should be excluded in the opinion of the investigator
7. Participation in another interventional clinical trial within 30 days of signing the Information and Consent Form (ICF)
8. Pregnant female patient

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female
2. Diagnosed with chronic stable heart failure
3. NYHA functional class II to ambulatory class IV
4. Peripheral oxygen saturation on fingertip pulse oximetry (SpO2) ≤96% at rest
5. Willingness and ability to use a POC and with no allergy to cannula material
6. Patient with the capacity to provide informed consent

Exclusion Criteria:

1. Contraindication to the use of POC
2. Patient currently hospitalized or requiring hospitalization
3. Current acute decompensated HF requiring augmented therapy with vasodilator agents, and/or inotropic drugs, and/or augmented therapy or i.v. therapy with diuretics
4. History of acute coronary syndrome (unstable angina or myocardial infarction) within 3 months prior to study enrollment
5. Patient unable to walk
6. Patient who should be excluded in the opinion of the investigator
7. Participation in another interventional clinical trial within 30 days of signing the Information and Consent Form (ICF)
8. Pregnant female patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Walking distance during the 6MWT | 6 minutes
  Walking distance during the 6MWT
Oxygen saturation | At 3 minutes (middle of the 6MWT)
  Oxygen saturation on fingertip pulse oximetry
Oxygen saturation | At 6 minutes (end of the 6MWT)
  Oxygen saturation on fingertip pulse oximetry
Oxygen saturation | At 9 minutes (3 minutes after the end of the 6MWT)
  Oxygen saturation on fingertip pulse oximetry
Heart rate | At 3 minutes (middle of the 6MWT)
  Heart rate
Heart rate | At 6 minutes (end of the 6MWT)
  Heart rate
Heart rate | At 9 minutes (3 minutes after the end of the 6MWT)
  Heart rate
Modified Borg Scale | At 3 minutes (middle of the 6MWT)
  Borg CR10 Scale (modified Borg Dyspnoea Scale). Scale with 0-10 scoring, where 0 means no Exertion and 10 means Maximal Exertion.
Modified Borg Scale | At 6 minutes (end of the 6MWT)
  Borg CR10 Scale (modified Borg Dyspnoea Scale). Scale with 0-10 scoring, where 0 means no Exertion and 10 means Maximal Exertion.
Modified Borg Scale | At 9 minutes (3 minutes after the end of the 6MWT)
  Borg CR10 Scale (modified Borg Dyspnoea Scale). Scale with 0-10 scoring, where 0 means no Exertion and 10 means Maximal Exertion.

SECONDARY OUTCOMES:
Adverse Events | Study period of approximately 5 hour on study day.
  Adverse events (AEs) and serious adverse events (SAEs)
Tolerance to POC | 6 minutes
  Ability (yes or no) to complete the 6MWT with the POC

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided